CLINICAL TRIAL: NCT00884247
Title: A Prospective, Non Interventional Study to Evaluate the Effects on Quality of Life, Symptoms and Productivity in Patients With Gastroesophageal Reflux Disease (GERD) After 6 Weeks Structured Treatment in a Company Health Care Setting
Brief Title: Structured Treatment of Gastroesophageal Reflux in a Company Health Care Setting, -Effect on Quality of Life, Symptoms and Productivity
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Svante Sjöstedt/MC MDOTA, AstraZeneca
Other Study IDs: NIS-GSE-DUM-2009/1
Record Dates: First submitted 2009-04-17; First posted 2009-04-20 (Estimated); Last update posted 2010-12-07 (Estimated); Status verified 2010-12

CONDITIONS: GERD
Keywords: GERD; Quality of life; Structured treatment
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The study aims to evaluate if a GERD treatment programme, in accordance with current regional recommendations, in a company health care setting, has an impact on health related quality of life (HRQoL), symptoms, and productivity in GERD patients.

ELIGIBILITY:
Inclusion Criteria:

* Female and/or male aged > 18 years
* Diagnosis of GERD confirmed
* Prescription of GERD treatment or already receiving GERD treatment

Exclusion Criteria:

* Any symptom suggesting a need for further investigation
* Previous participation in the present study
* Current participation in a clinical study or participation in a clinical study during the last 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Company health care setting
Sampling Method: Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2009-04; Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Svante Sjöstedt, MD, PhD, Study Director — AstraZeneca Sweden; Dan Regberg, MD, Principal Investigator — AstraZeneca Sweden
Locations (1):
- Research Site, Hälsocenter, Södertälje, Sweden